CLINICAL TRIAL: NCT02159924
Title: Posture and Mobility Measurements of the Upper Quadrant in Asymptomatic Subjects by Means of a Smartphone
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Nuno Morais, Master student in traditional chinese medicine, Universidade do Porto
Other Study IDs: ROM_iPhone_2014
Record Dates: First submitted 2014-06-01; First posted 2014-06-10 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Posture and Mobility of the Upper Quadrant
Keywords: Smartphone measurements; Orientation; Range of motion; Median nerve neurodynamic test; Posture; Thoracic spine; Shoulder girdle
MeSH Terms: conditions — Orientation, Spatial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Asymptomatic

SUMMARY:
This study aims to investigate posture-mobility associations in the upper quadrant by means of smartphone measurements

DETAILED DESCRIPTION:
One purpose of this study is to measure the magnitude of the thoracic kyphosis, thoracic spine extension, and side-to-side differences in scapular protraction and elbow extension range of motion during the median nerve neurodynamic test through a smartphone (iPhone 4, app Compass, iOS 7.1.1), and to assess the intrarater agreement parameters.

Another purpose is to assess associations between thoracic kyphosis, thoracic spine extension, scapular protraction and the resting length of the pectoralis minor muscle through smartphone, photographs and tape measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Normal mobility in the joints of the upper quadrant

Exclusion Criteria:

* complaints in the upper quadrant over the past 3 months
* significant deformities in the upper quadrant
* leg length discrepancy > 1.5 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomatic subjects from scholar community
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Elbow extension range of motion | At the time of the assessment
  Elbow extension range of motion (in degrees) during the median nerve neurodynamic test is measured by means of a smartphone (iPhone 4, app Compass, iOS 7.1.1)
Thoracic kyphosis orientation | At the time of the assessment
  The magnitude of the thoracic kyphosis (in degrees) in the standing upright position is measured by means of a smartphone (iPhone 4, app Compass, iOS 7.1.1)
Thoracic spine extension range of motion | At the time of the assessment
  The extension range of motion of the thoracic spine (in degrees) in the standing upright position is measured by means of a smartphone (iPhone 4, app Compass, iOS 7.1.1)
Scapular protraction orientation | At the time of the assessment
  The magnitude of the scapular protraction (in degrees) in the standing upright position with the arms at rest is measured by means of a smartphone (iPhone 4, app Compass, iOS 7.1.1)
Pectoralis minor muscle resting length | At the time of the assessment
  Pectoralis minor muscle resting length (in centimeters) with the arms at rest is measured by means of a measuring tape in the standing upright position
Thoracic kyphosis orientation | At the time of the assessment
  The magnitude of the thoracic kyphosis (in degrees) in the standing upright position is measured on digital photographs by means of a computer software
Thoracic spine extension range of motion | At the time of the assessment
  The extension range of motion of the thoracic spine (in degrees) in the standing upright position is measured on digital photographs by means of a computer software

CONTACTS AND LOCATIONS:
Overall Officials: Nuno V Morais, MSc, Principal Investigator — Instituto Politécnico de Leiria
Locations (1):
- Escola Superior de Saúde do Instituto Politécnico de Leiria, Leiria, Leiria District, Portugal

REFERENCES:
- [Derived] Cruz J, Morais N. Intrarater Agreement of Elbow Extension Range of Motion in the Upper Limb Neurodynamic Test 1 Using a Smartphone Application. Arch Phys Med Rehabil. 2016 Nov;97(11):1880-1886. doi: 10.1016/j.apmr.2016.05.001. Epub 2016 May 17. PMID 27207436